CLINICAL TRIAL: NCT05386498
Title: Comparison of Proximal Contacts and Contours in Class II Composite Restoration With Pre-cured Composite Inserts Versus Contact Making Instrument Technique. A Randomized Control Clinical Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUI/CTR/2022/7
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Class 2 Dental Cavity

STUDY DESIGN:
Intervention Model Description: The study is a single centre based randomized control trial where the intervention arm 1 will get their class 2 restorations done with precured composte insert technique.
  The intervention arm 2 will recieve treatment with contact making instrument technique.
  The intervention arm 3 patients will be the control group and will recieve treatment of their class 2 restoration with the incremental composite layering techique. The study will be conducted on patients seeking class 2 restorations at the operative department of foundation university college of dentistry. Allocation of the patients in treatment groups will be done by simple randomization using the lottery method.
Who Masked: Participant, Outcomes Assessor
Masking Description: Two consultants will be assessors who will be calibrated by demonstration of outcome assessment.
  Series of assessments will be done on patients and inter assessor reliability will be determined.
  An agreement of 0.7 by intraclass correlation coeffiecient will be considered as good reliability.
  At the time of treatment a single assessor out of the two, will be blinded to the treatment allocation and will check the contact tightness of the filling. Masking will be ensured as the assessors will not be present at the time of treatment allocation or at the time of treatment administration and will be involved only once the procedure is complete. Assessment will be done using a waxed floss passed between the filling and the adjacent tooth. Due to interventional nature of the study the treating dentist cannot be blinded to the allocation of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Precure composite insert technique (Experimental): After curing of bonding agent a 2mm increment of composite will be placed on the gingival floor of the cavity and cured. a measured volume of composite(3mm height and 2mm width) will be cured outside the oral cavity on a flat plastic instrument for 40 seconds. a second increment of composite will be placed on the cavity and the precured composite will be pressed in the uncured increment and pressed outward against the matrix band and light cured for 20 seconds the rest of the cavity will be filled using the oblique layering technique.
  Interventions: Procedure: precured composite insert technique
- Contact Making Instrument (Experimental): a 1-2mm increment of the composite will be placed in the gingival floor of the proxial box.
  a contact forming instrument will be placed in this uncured increment and an outward force will be applied using the instrument from the inside of the matrix band. The composite will then be cured for 20 seconds to achieve a tight contact.
  Interventions: Procedure: Contact making instrument
- Incremental composite layering technique (Active Comparator): Increments will be placed in 1-2mm increments in oblique layering manner by a flat plastic instrument and condenser .Each increment will be cured for 20 seconds till the cavity is slightly overfilled.
  Interventions: Procedure: Incremental composite layering technique

INTERVENTIONS:
Procedure: precured composite insert technique — After curing of bonding agent a 2mm increment of composite will be placed on the gingival floor of the cavity and cured. a measured volume of composite(3mm height and 2mm width) will be cured outside the oral cavity on a flat plastic instrument for 40 seconds. a second increment of composite will be placed on the cavity and the precured composite will be pressed in the uncured increment and pressed outward against the matrix band and light cured for 20 seconds the rest of the cavity will be filled using the oblique layering technique.
  Arms: Precure composite insert technique
Procedure: Contact making instrument — a 1-2mm increment of the composite will be placed in the gingival floor of the proxial box.
  a contact forming instrument will be placed in this uncured increment and an outward force will be applied using the instrument from the inside of the matrix band. The composite will then be cured for 20 seconds to achieve a tight contact.
  Arms: Contact Making Instrument
Procedure: Incremental composite layering technique — Increments will be placed in 1-2mm increments in oblique layering manner by a flat plastic instrument and condenser .Each increment will be cured for 20 seconds till the cavity is slightly overfilled.
  Arms: Incremental composite layering technique

SUMMARY:
The objective of this randomized control cinical trial will be to compare the effectiveness of precured composite inserts in obtaining tight and adequate conatacts in class 2 restorations when compared with the contact making instrument technique among patients treated at the operative depatment of Foundation Umiversity College of Dentistry.

This is a single centre based randomized control clinical trial in which intervention arm 1 will get there class 2 restoration done with precured composite inserts and interention arm 2 will recieve treatment with contact making instrument technique. The control arm will recieve restoration using the conventional composite layering technique.

DETAILED DESCRIPTION:
Study design : randomized control clinical trial with three intervention arms

Study setting : operative department , foundation university college of dentistry Islamabad Pakistan.

Sample size : the sample size was calculated using the NCSS PASS software. A total od 180 patients will be tested in the study divided in three groups of 60 patients each. Consent will be taken from pateints on a standardized form approved by the ethics review committe in the operatory where the initial assessment will be done.

Procedure:

1. number of operaters will be restricted two, with similar level of experience in order to minimize operater variation
2. the investigator and co investigator will calibrate each other on the sequence of the procedure and assessment to enhance standardization of procedure
3. local anaesthesia will be given to patients using lidocaine 2% solution available for dental use in 1.8 ml carpule
4. rubber dam will used for isolation and moisture control in the working field.
5. the tooth to be restored will be seperated from the adjacent tooth using wooden wedges.this will allow seperation of teeth.
6. cavity preparation will be done using a high speed handpiece(W&H) with a round bur(prima) (no1/6 or 1/4). After initial penetration through enamel the carious lesion will be excavated using a a carbide bur in a slow speed handpiece.

   after caries removal any unsupported enamel at the gingival floor will be removed using a gingival margin trimmer.

   the cavity shape will be finalized using a pear shaped bur(243).
7. the width of the final cavity will be measured using a perio probe from the buccal or labial cavo surface margin. Only cavities with less than 1/2 the width of the distance or less from the buccal or lingual cusp tip will be included in the study.
8. sectional metal matrix (unimatrix by TDV Brazil,1/4" by 0.0015,1/4" by.002,height and thickness of matrix) will be applied after removing the previously placed wooden wedges. The wedges will be reintroduced after sectional matrix application.
9. the cavity will be etched using 37% phosphoric acid etchant(30 seconds enamel and 15 seconds dentine) followed by rinsing for 30 seconds with the triple syringe. the cavity will be gently air dried while keep a dried cotton pellet in the cavity to absorb excess moisure for 30 to 45 seconds.Prime and Bond NT (Dentsply) adhesive will be applied to the cavity followed by curing for 20 seconds with an led based curing light (O-light,DTE wavelength of 400nm visible blue light). The cavities in all intervention arms will be restored with neo spectre NT composite(dentsply). (the detail of each intervention arm is given under their respective headings)
10. after the cavities are filled the matrix band and the wedges will be removed.the cavity will be finished using diamond burs and composite finishing spirals(azdent). occlusal adjustment will be done where needed using articulating paper.
11. the final restoration will be polished using diamond polishing paste(ultradent) and goat hair brushes (ultradent)

Assessment

1. assessment will be done by passing waxed dental floss between the filling and adjacent tooth by a single independent assessor blinded to the treatment allocation.
2. outcome will be assessed using the contact tightness and contour component of the modified USPHS rating scale
3. data collection will be done at the end of the treatment using a printed porforma for recording the study variables.

Data analysis

1. will be done using spss 26
2. for continouse variables like age and cavity wifth and depth , mean and standard deviations will be computed.

   comparison of these variable will be done by one way anova test
3. for categorical variables like gender, type of tooth,location of cavity,contact tightness and contour(outcome variables) frequencies in percentages will be reported. these variables will be compared using kruskal-wallis test at 0.05 level of significance

ELIGIBILITY:
Inclusion criteria

1. patient requiring treatment for class 2 cavity
2. patient age 12 to 55 years
3. Maxillary and Mandibular first and second premolar
4. Maxillary and Mandibular first and second molar
5. Maximum occlusal cavo surface width of 2/3rd of intercuspal width
6. Cavity depth upto 3/4th of occlusocervical length measured from diagnostic radiograph
7. Teeth with adjacent fully erupted teeth adjacent to a cavity side Exclusion criteria

1)Mentally and physically handicapped patient 2)Pregnant females 3)Patients with naturally spaced teeth 4)Patients with moderate or advanced periodontitis 5)Endodontically treated teeth 6)Teeth with excessive occlusal wear and erosion of teeth 7)Tooth adjacent to cavity side is missing 8)Teeth with orhtodontic bands and brackets 9)Tooth adjacent to cavity side is restored

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-03-30 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Contact tightness and Contour of Class 2 composite restoration | 1 day
  The contact tightness and contour of the filling will be assessed using the modified united states public health service system rating scale which has is used in studies on dental materials.